CLINICAL TRIAL: NCT04508699
Title: Semantic Learning Deficits in School Age Children With Developmental Language Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Alyson Abel Mills, Associate Professor, San Diego State University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: R21DC018865 (NIH)
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Developmental Language Disorder
Keywords: Semantic Learning; ERP; N400; ERSP
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Intervention Model Description: Compare behavioral and EEG outcomes of semantic learning in children with and without developmental language disorder
Who Masked: Participant, Care Provider
Masking Description: Some participants and care providers might not be aware of their child's language impairment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Developmental language disorder (Experimental): Children with language impairment but in the absence of cognitive deficits
  Interventions: Other: semantic learning
- Typical language (Active Comparator): Children with typical language development and typical cognitive development
  Interventions: Other: semantic learning

INTERVENTIONS:
Other: semantic learning — Experimental semantic learning from linguistic context task

SUMMARY:
School age children with developmental language disorder (DLD) have known semantic learning deficits but what is less well understood is why semantic learning is difficult for these children. This project will combine behavioral and brain methods to investigate the cognitive and linguistic processes underlying semantic learning in children with DLD compared to typically developing peers. The outcomes will have implications for semantic learning intervention approaches in DLD.

DETAILED DESCRIPTION:
This project will elucidate deficits in learning semantic information in developmental language disorder (DLD, formerly referred to as specific language impairment) by combining behavioral and neural measures to examine differences in the semantic learning process between school-age children with and without DLD. Vocabulary knowledge, particularly semantic knowledge, has a critical influence on reading comprehension and academic success. Despite the strong association between vocabulary knowledge and academic success, vocabulary is an under-recognized area of deficit in school-age children with DLD. Younger children with DLD have well-established deficits in vocabulary and word learning and weaknesses in semantic knowledge. Additionally, the rate of vocabulary growth in children with DLD decreases compared to typically developing peers around age 10 and semantic representations of known vocabulary items are sparse. Even with this knowledge, the field's ability to make progress toward improved semantic learning in school age DLD is hindered by the lack of basic information on the underlying nature of the semantic learning deficits in this population. This project establishes how and why semantic learning differs between school-age children with and without DLD, providing a much-needed theoretical foundation for clinical research.

Storkel, expanding on an adult word learning model by Leach and Samuel, provides a clearly testable account of word learning that has been used with children with DLD. This account involves three processes: 1) triggering, in which a new lexical encounter is compared to existing lexical representations, 2) configuration, which adds information to the expanding lexical representation, and 3) engagement, which examines how the new lexical representation behaves dynamically with existing representations. The configuration process is arguably the most critical for semantic development. Successful configuration requires the simultaneous engagement of cognitive and linguistic processes, such as attention, inhibition, working memory, and semantic and syntactic processing. While it is widely accepted that configuration is the most affected word learning process in DLD, what is unknown is what underlies deficits in configuration and whether these deficits vary across the DLD profile. These questions are further compounded by difficulty measuring configuration and associated processes, given that they are largely internal, and therefore invisible. Electroencephalography (EEG) addresses this invisibility problem by allowing for a real-time examination of unconscious levels of semantic learning and cognitive and linguistic processes. A combined EEG-behavioral methods approach can illustrate how children with DLD are approaching configuration in terms of the relative contribution of these processes. The central hypothesis of this research is that children with DLD engage cognitive and linguistic processes at different points during configuration compared to their typical peers, resulting in poorer semantic learning outcomes.

To test the central hypothesis, the investigators will record behavioral and EEG data from 10-12 year old children with DLD and typical-language peers as they complete a semantic learning task. This age aligns with the point where vocabulary growth rates in DLD further diverge from typical peers [6]. In the semantic learning task, children listen to sets of three sentences that all end with the same nonword: half of the sentence triplets support learning meaning of the nonword, half do not. The investigators will analyze EEG data for event-related potentials (ERPs) as well as changes in neural oscillations (time frequency analysis). The investigators will combine EEG and behavioral measures to examine the following aims:

Aim 1. To investigate the cognitive and linguistic processes underlying configuration in children with DLD and typical language (TL) peers. This aim will include data from the semantic learning task. Based on the assessment of behavioral outcomes, the investigators predict that the TL group will be more accurate in semantic learning than the DLD group. ERP analyses will focus on the N400 component, associated with semantic processing. Time frequency analysis will focus on changes in the theta (4-8 Hz) and alpha (8-12 Hz) frequency bands, typically associated with lexical retrieval and attention/inhibition, respectively. For both neural measures, the investigators predict engagement of the same components (N400, theta, alpha) across groups but different patterns of change in those components during configuration between groups.

Aim 2. To investigate individual differences in configuration in children with DLD and TL peers. This aim will include data from the semantic learning task and a behavioral assessment battery. Assessment of behavioral data will focus the types of errors children make during semantic learning. The investigators expect that children with DLD will provide incorrect meanings for the nonword that best fit with the first sentence in the triplet and that TL children will provide incorrect meanings that best fit with the last sentence. The investigators will also examine individual differences related to semantic learning outcomes and fine-grained differences in N400 learning effects across groups. Here, the investigators expect that individual differences in general language ability and semantic knowledge, measured via the behavioral assessment battery, will be most predictive of both behavioral semantic learning and N400 change during learning.

ELIGIBILITY:
Inclusion Criteria:

* history of typical language development or history of language or literacy difficulties
* must be willing to wear EEG cap
* must be able to sit still for 1.5 hours to complete experimental tasks
* must be literate

Exclusion Criteria:

* neurological disorders (i.e., ASD, ADHD)
* significant neurological history (i.e., head injury, epilepsy)
* left handedness
* primary language other than English
* medication other than over-the-counter allergy medications
* and/or nonverbal IQ less than 70

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 167 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alyson Abel, PhD, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from online sources (e.g., Craiglist, Facebook groups), word of mouth, clinical sites (on-campus Clinic, private clinics), local public schools, and the local University.
Pre-assignment Details: No events to report.
Groups:
- Typical Language Children: Children with typical language development and typical cognitive development
Period: Overall Study
Arm/Group | Developmental Language Disorder | Typical Language Children
Started | 15 | 97
Completed | 13 | 80
Not Completed | 2 | 17
Not completed — Lack of Efficacy | 2 | 15
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Developmental Language Disorder | Typical Language Children | Total
Number analyzed (Participants) | 15 | 97 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 97 | 112
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10 (1.69) | 11.7 (2.53) | 11.54 (2.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 50 | 55
  Male | 10 | 47 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 14 | 18
  Not Hispanic or Latino | 4 | 39 | 43
  Unknown or Not Reported | 7 | 44 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 7 | 7
  White | 4 | 24 | 28
  More than one race | 3 | 13 | 16
  Unknown or Not Reported | 8 | 49 | 57
Region of Enrollment [Number; unit: participants]
  United States | 15 | 97 | 112

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Correct Semantic Meaning Identification
Description: Accuracy on the semantic learning task. Did they correctly identify when there was a meaning or did they say there was no meaning when there should have been one (incorrect response) Higher is better outcome
Time Frame: immediately following treatment, on the same day as treatment, within 30 minutes
Population: Data analyzed from complete data sets
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Developmental Language Disorder | Typical Language Children
Number analyzed (Participants) | 15 | 87
percentage of correct responses
  Meaning condition accuracy | 73.6 (16.4) | 75.12 (14.7)
  No meaning condition accuracy | 77.1 (19.5) | 82.3 (15.2)
Statistical Analysis 1: Comparison: Developmental Language Disorder vs Typical Language Children; Test type: Other; p = 0.36, t-test, 1 sided

2. Primary Outcome: N400 Amplitude - Sentence 1
Description: Mean amplitude (measured in microvolts) of the N400 time locked to the target word in sentence 1 collapsed across groups matched for age. Meaning plus condition only.
  Smaller/more negative indicates more effortful (harder) processing and larger/more positive indicates less effortful (easier) processing.
Time Frame: immediately following treatment, on the same day as treatment, within 30 minutes
Population: Children with usable EEG data and matched for age
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Developmental Language Disorder | Typical Language
Number analyzed (Participants) | 14 | 14
microvolts | -.1 (.002) | -.27 (.0045)
Statistical Analysis 1: Comparison: Developmental Language Disorder vs Typical Language; Test type: Other; p < 0.05, ANOVA — reported p-value was calculated, is not indicating the threshold for statistical significance

3. Primary Outcome: Theta Changes
Description: Changes in theta band activity (measured in hertz) from sentence 1 to sentence 3, time locked to the final word in the sentence.
  Smaller/more negative indicates more effortful (harder) processing and larger/more positive indicates less effortful (easier) processing.
Time Frame: immediately following treatment, on the same day as treatment, within 30 minutes
Population: Participants with complete EEG datasets, age matched
Measure: Mean (Standard Deviation); unit: Hertz
Arm/Group | Developmental Language Disorder | Typical Language
Number analyzed (Participants) | 11 | 11
Hertz | .0521 (.478) | .121 (.21)
Statistical Analysis 1: Comparison: Developmental Language Disorder vs Typical Language; Test type: Other; p < 0.05, ANOVA — reported p-value was calculated, is not indicating the threshold for statistical significance

4. Primary Outcome: N400 Amplitude - Sentence 2
Description: Mean amplitude (measured in microvolts) of the N400 time locked to the target word in sentence 2 collapsed across groups matched for age. Meaning plus condition only.
  Smaller/more negative indicates more effortful (harder) processing and larger/more positive indicates less effortful (easier) processing.
Time Frame: immediately following treatment, on the same day as treatment, within 30 minutes
Population: Participants with usable EEG data, groups matched for age
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Developmental Language Disorder | Typical Language
Number analyzed (Participants) | 14 | 14
microvolts | -0.1 (0.005) | 0.075 (0.003)
Statistical Analysis 1: Comparison: Developmental Language Disorder vs Typical Language; Test type: Other; p < 0.05, ANOVA — reported p-value was calculated, is not indicating the threshold for statistical significance

5. Primary Outcome: N400 Amplitude - Sentence 3
Description: Mean amplitude (measured in microvolts) of the N400 time locked to the target word in sentence 3 collapsed across groups matched for age. Meaning plus condition only.
  Smaller/more negative indicates more effortful (harder) processing and larger/more positive indicates less effortful (easier) processing.
Time Frame: immediately following treatment, on the same day as treatment, within 30 minutes
Population: Children with usable EEG data and matched for age
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Developmental Language Disorder | Typical Language
Number analyzed (Participants) | 14 | 14
microvolts | 0.221 (.004) | .662 (0.07)
Statistical Analysis 1: Comparison: Developmental Language Disorder vs Typical Language; Test type: Other; p < 0.05, ANOVA — reported p-value was calculated, is not indicating the threshold for statistical significance

6. Secondary Outcome: General Language Level
Description: Full measure title: Clinical Evaluation of Language Fundamentals - 5th edition Standardized language omnibus measure Raw scores converted to t-score: 100 indicates population mean and standard deviation is 15 Higher scores indicate a better outcome and lower scores indicate a poorer outcome Typical range = 85-115; below 80 is considered in the sub-clinical range indicating the presence of a language disorder
Time Frame: baseline
Population: Data analyzed from complete datasets
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Developmental Language Disorder | Typical Language Children
Number analyzed (Participants) | 15 | 92
t-score | 73.2 (11.6) | 110.9 (11.86)
Statistical Analysis 1: Comparison: Developmental Language Disorder vs Typical Language Children; Test type: Other; p < 0.00001, t-test, 1 sided — reported p-value was calculated, is not indicating the threshold for statistical significance

7. Secondary Outcome: Nonverbal Cognition
Description: Full measure title: Wechsler Intelligence Scale for Children - 5th edition Nonverbal index subtests administered, considered the nonverbal subscale For the nonverbal subscale, raw scores converted to t-score: 100 indicates population mean and standard deviation is 15 Higher scores indicate a better outcome and lower scores indicate a poorer outcome Typical range = 85-115; below 70 is considered in the sub-clinical range indicating the presence of intellectual disability
Time Frame: baseline
Population: Participants with completed data sets
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Developmental Language Disorder | Typical Language Children
Number analyzed (Participants) | 15 | 92
T-score | 86.2 (11.2) | 106.93 (12.3)
Statistical Analysis 1: Comparison: Developmental Language Disorder vs Typical Language Children; Test type: Other; p < 0.00001, t-test, 1 sided — reported p-value was calculated, is not indicating the threshold for statistical significance

8. Secondary Outcome: Nonword Repetition Task
Description: experimental task gauging phonological memory
Time Frame: baseline
Population: Participants with complete datasets
Measure: Mean (Standard Deviation); unit: percent consonants correct
Arm/Group | Developmental Language Disorder | Typical Language Children
Number analyzed (Participants) | 15 | 94
percent consonants correct | 83.9 (9.6) | 92.9 (5.3)
Statistical Analysis 1: Comparison: Developmental Language Disorder vs Typical Language Children; Test type: Other; p < 0.00001, t-test, 1 sided — reported p-value was calculated, is not indicating the threshold for statistical significance

ADVERSE EVENTS:
Time Frame: 4 hour data collection for each participant
Arm/Group | Developmental Language Disorder | Typical Language Children
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/97
Other Adverse Events (participants affected / at risk) | 0/15 | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT04508699/Prot_SAP_000.pdf